CLINICAL TRIAL: NCT06609902
Title: Future Self: An Episodic Future Thinking Intervention for Comorbid Tobacco Use Disorder and Bipolar Disorder
Brief Title: A Future Thinking Intervention for Comorbid Tobacco Use Disorder and Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexandra K. Gold, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024P000546
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Bipolar Disorder; Tobacco Use Disorder
Keywords: bipolar disorder; comorbid tobacco use disorder; smoking cessation
MeSH Terms: conditions — Bipolar Disorder; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: This is a treatment development study that begins with an open non-randomized pilot trial (N = 10) in which we will test the manual developed for Future Self-BD by assessing the acceptability and feasibility of Future Self-BD. After completion of the non-randomized pilot trial and subsequent revisions to the Future Self-BD manual, we will conduct a parallel randomized controlled trial comparing Future Self-BD (N = 30) to a control treatment, Daily Check-Ins (N = 30). Future Self-BD and Daily Check-Ins involve six, weekly, 1.5-2 hour sessions and one 1.5 hour follow-up session one month after completion of the sixth session
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Future Self-BD (Experimental): Experimental Arm utilizing the Future Self-BD Intervention.The Future Self group will attend 6 virtual sessions during which they will be encouraged to vividly generate personal and positive future events that they anticipate may be benefited by smoking cessation. All participants will complete the adjusting amount discounting task. All participants will also receive brief, CBT-based smoking cessation counseling. This group will involve one follow-up session one month after the sixth session. Each session will be conducted on HIPAA-compliant Zoom and led by the PI, Dr. Gold.
  Interventions: Behavioral: Future Self-BD
- Daily Check-Ins (Active Comparator): Active comparator arm utilizing Daily Check-Ins (DCI). The DCI group will attend 6 virtual sessions during which they will complete the adjusting amount discounting task and receive brief, CBT-based smoking cessation counseling (consistent with counseling received by Future Self-BD). This group will involve one follow-up session one month after the sixth session. Each session will be conducted on HIPAA-compliant Zoom and led by the PI, Dr. Gold.
  Interventions: Behavioral: Daily Check-Ins

INTERVENTIONS:
Behavioral: Future Self-BD — The Future Self group will attend 6 virtual sessions during which they will be encouraged to vividly generate personal and positive future events that they anticipate may be benefited by smoking cessation. All participants will complete the adjusting amount discounting task. All participants will also receive brief, CBT-based smoking cessation counseling. This group will involve one follow-up session one month after the sixth session. Each session will be conducted on HIPAA-compliant Zoom and led by the PI, Dr. Gold.
  Arms: Future Self-BD
Behavioral: Daily Check-Ins — The Daily Check-Ins (DCI) group will attend 6 virtual sessions during which they will complete the adjusting amount discounting task and receive brief, CBT-based smoking cessation counseling (consistent with counseling received by Future Self-BD). This group will involve one follow-up session one month after the sixth session. Each session will be conducted on HIPAA-compliant Zoom and led by the PI, Dr. Gold.
  Arms: Daily Check-Ins

SUMMARY:
Future Self-BD is a 6-session virtual intervention that encourages participants to vividly generate personal and positive future events that they anticipate may be benefited by smoking cessation. Each session will be conducted on HIPAA-compliant Zoom and led by the PI (Dr. Gold).

DETAILED DESCRIPTION:
This is a treatment development study that begins with an open non-randomized pilot trial (N = 10) in which we will test the manual developed for Future Self-BD by assessing the acceptability and feasibility of Future Self-BD. After completion of the non-randomized pilot trial and subsequent revisions to the Future Self-BD manual, we will conduct a parallel randomized controlled trial comparing Future Self-BD (N = 30) to a control treatment, Daily Check-Ins (N = 30). Future Self-BD and Daily Check-Ins involve six, weekly, 1.5-2 hour sessions and one 1.5 hour follow-up session one month after completion of the sixth session; thus, participants will be enrolled in the study for a period of 10 weeks. Assessments will occur at all study sessions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older
* Have a diagnosis of BD I or II
* Have a diagnosis of tobacco use disorder
* Be engaged in outpatient treatment with a medical provider
* Be on a stable dose of a mood-stabilizing medication
* Smoke an average of at least 5 cigarettes per day for the past 30 days at baseline (based on the Heaviness of Smoking Index(Heatherton et al., 1989))
* Be interested in quitting smoking
* Not currently or in the past 3 months be receiving smoking cessation treatment.

Exclusion Criteria:

* Current psychosis
* Intent to harm oneself with an associated plan and intent to act on suicidal thoughts
* Experiencing severe symptoms of depression and/or hypomania that may warrant a higher level of care (a Patient Health Questionnaire-9 total score ≥ 20(Kroenke et al., 2001) and/or an Altman Self-Rating Mania Scale total score ≥ 6(Altman et al., 1997) will trigger further clinician evaluation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the Study Intervention | Week: 6
  The Client Satisfaction Questionnaire (CSQ-8) will be administered at the end of session 6 to assess intervention acceptability via participant satisfaction with the intervention, with higher scores reflecting more satisfaction
Feasibility of the Study Intervention | Week: 6
  We will assess feasibility via the frequency of participants who attend session 6 (i.e., retention).
Feasibility of the Study Intervention | Week: 6
  We will assess feasibility via the frequency of participants who complete greater than or equal to 75% of cue recalls (Future Self-BD) or open-ended questions (Daily Check-Ins) and coach-led sessions (i.e.,completion).

SECONDARY OUTCOMES:
Self-Efficacy to Resist Smoking as Assessed by the Smoking Self-Efficacy Questionnaire(SEQ-12) | Week: 1, 6, 10
  Participant self-efficacy to resist smoking will be assessed by the Smoking Self-Efficacy Questionnaire (SEQ-12) to assess how confident someone is that they will be able to resist smoking across various situations. It will be administered at sessions 1, 6, and follow-up.
Participant Motivation to Quit Smoking | Week: 1, 6, 10
  Participant motivation to quit smoking will be assessed using a single item that asks participants to rate how motivated they are to quit smoking on a scale from 0 (not at all motivated) to 10 (extremely motivated). It will be administered at sessions 1, 6, and follow-up.
Seeking Smoking Cessation Treatment as Assessed by The Seeking Smoking Cessation Treatment Questionnaire | Week: 1, 2, 3, 4, 5, 6, 10
  The Seeking Smoking Cessation Treatment Questionnaire will be administered at sessions 1-6 and follow-up. This questionnaire assesses whether participants sought smoking cessation treatment since the last session, the nature of this treatment (i.e., NRT), how they sought this treatment, and whether they are interested in receiving a referral for smoking cessation treatment at the day's session.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra K Gold, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States